CLINICAL TRIAL: NCT06949956
Title: Administration of Fingolimod in Greek Patients With Multiple Sclerosis for the Evaluation of the Efficacy and Safety, Based on the Standard Clinical Practice.
Brief Title: Administration of Fingolimod in Greek Patients With Multiple Sclerosis.
Acronym: FILYRA
Status: Not yet recruiting | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Collaborators: AHEPA University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-FIN-EL-152
Record Dates: First submitted 2025-04-28; First posted 2025-04-29 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: RRMS; ARR; EDSS; Fingolimod
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis patients: Multiple Sclerosis patients already receiving fingolimod and who have available follow-up data for at least 12 months prior to study entry, sufficient to calculate the annualized relapse rate.

SUMMARY:
The goal of this observational study is to evaluate the efficacy of fingolimod through the estimation of the annualized relapse rate (ARR) over a period of 2 years.

Participants who are already taking fingolimod as part of their regular medical care for MS will answer questions about their medical history for the past 1 year and for their status for the next 2 years.

DETAILED DESCRIPTION:
The efficacy of fingolimod will be assessed:

* by calculating the difference in annualized relapse rate (ARR) between the 12-month period prior to study entry and that which will occur during the study at 0, 6, 12, 18 and 24 months of treatment
* by calculating the change in EDSS score between the 12-month period prior to study entry and that which will occur during the study at 0, 6, 12, 18 and 24 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 18 years of age.
2. Consent and compliance of participants with the treatments and procedures of the study.
3. Patients diagnosed with relapsing-remitting multiple sclerosis (RRMS) according to the revised McDonald 2017 criteria.
4. Patients who are receiving fingolimod, according to the drug's Summary of product Characteristics (SmPC).
5. Patients with available follow-up data for at least 12 months prior to their inclusion in the study, which are sufficient to calculate the annualized relapse rate.

Exclusion Criteria:

1. Patients under 18 years of age.
2. Patients with a contraindication to taking fingolimod according to the drug's Summary of product Characteristics (SmPC).
3. Patients with a history of mental illness, substance abuse, to a degree that may prevent their participation in the study.
4. Patients participating in another research protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll patients with relapsing-remitting multiple sclerosis (RRMS) who are already receiving the active substance fingolimod.
  Patients must have at least 12 months of follow-up data available prior to study entry, sufficient to calculate the annualized relapse rate.
  No additional diagnostic or monitoring procedures will be required for patient participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate, ARR | 2 years
  The difference in the annualized relapse rate (ARR) between the twelve-month period prior to study entry and that which will occur during the study.

SECONDARY OUTCOMES:
Expanded Disability Status Scale, EDSS | 2 years
  The change in Expanded Disability Status Scale (EDSS) score between the 12-month period before study entry and during the study. EDSS scale provides a score ranging from 0 to 10, where lower scores indicate less disability and higher scores indicate greater disability.
Progression Independent of Relapse Activity, PIRA | 2 years
  Assessment of patients with Progression Independent of Relapse Activity (PIRA), through the roving EDSS method.
Further calculation of Progression Independent of Relapse Activity (PIRA) taking into account clinical and imaging data (if available). | 2 years
  Further calculation of Progression Independent of Relapse Activity (PIRA) taking into account clinical data (SDMT, 9 Hole Peg-Test, Timed 25-Foot Walk tests) and imaging data (new/enlarging or enhancing lesions on Magnetic Resonance Imaging MRI, if available).
Quality of Life (QoL) of patients with multiple sclerosis. | 2 years
  Evaluation of Multiple Sclerosis International Quality of Life (MusiQoL) questionnaire scores at 0, 12 and 24 months of treatment. MusiQoL questionnaire have responses describing frequency/extent of an event on a five-point scale ranging from 'never/not at all' (option'1') to 'always/very much' (option '5').
Safety evaluation of the drug throughout the treatment period. | 2 years
  Recording of adverse events (AE) during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Grigoriadis, MD, Principal Investigator — AHEPA University Hospital of Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] Walton C, King R, Rechtman L, Kaye W, Leray E, Marrie RA, Robertson N, La Rocca N, Uitdehaag B, van der Mei I, Wallin M, Helme A, Angood Napier C, Rijke N, Baneke P. Rising prevalence of multiple sclerosis worldwide: Insights from the Atlas of MS, third edition. Mult Scler. 2020 Dec;26(14):1816-1821. doi: 10.1177/1352458520970841. Epub 2020 Nov 11. PMID 33174475
- [Background] Bakirtzis C, Grigoriadou E, Boziki MK, Kesidou E, Siafis S, Moysiadis T, Tsakona D, Thireos E, Nikolaidis I, Pourzitaki C, Kouvelas D, Papazisis G, Tsalikakis D, Grigoriadis N. The Administrative Prevalence of Multiple Sclerosis in Greece on the Basis of a Nationwide Prescription Database. Front Neurol. 2020 Sep 29;11:1012. doi: 10.3389/fneur.2020.01012. eCollection 2020. PMID 33132996